CLINICAL TRIAL: NCT00141336
Title: Pregabalin BID Open-Label Add-On Trial: An Open-Label, Multicenter Follow-On Study to Determine Long-Term Safety and Efficacy in Patients With Partial Seizures.
Brief Title: To Evaluate the Long-Term Safety and Efficacy of Pregabalin in Patients With Partial Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-035
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-01-01 (Estimated); Status verified 2006-12

CONDITIONS: Seizure Disorder, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To evaluate the long-term safety and tolerability of pregabalin in patients with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for preceding double-blind study
* Have received double-blind study medication and wish to receive open-label pregabalin.

Exclusion Criteria:

* Cannot have absence seizures

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750
Dates: Start 1999-11; Study Completion 2005-07

PRIMARY OUTCOMES:
Safety Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (79):
- United States (74):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Bakersfield, California
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Concord, California
  - Pfizer Investigational Site, Covina, California
  - Pfizer Investigational Site, El Cajon, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Marina Del Ray, California
  - Pfizer Investigational Site, Martinez, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Pinole, California
  - Pfizer Investigational Site, Redondo Beach, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, Danbury, Connecticut
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Ruston, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Golden Valley, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Concord, New Hampshire
  - Pfizer Investigational Site, Dover, New Hampshire
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Ridgewood, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Ridley Park, Pennsylvania
  - Pfizer Investigational Site, Upland, Pennsylvania
  - Pfizer Investigational Site, Cranston, Rhode Island
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Alexandria, Virginia
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Roanoke, Virginia
  - Pfizer Investigational Site, Sterling, Virginia
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Friday Harbor, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Morgantown, West Virginia
  - Pfizer Investigational Site, Marshfield, Wisconsin
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Canada (5):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario